CLINICAL TRIAL: NCT05419401
Title: A Phase I Study to Investigate the Absolute Bioavailability, Absorption, Metabolism, Distribution and Excretion of [14C]AZD5363 (Capivasertib) in Healthy Male Subjects
Brief Title: A Study to Investigate the Absolute Bioavailability, Absorption, Metabolism, Distribution and Excretion of [14C]AZD5363 (Capivasertib)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3614C00007
Record Dates: First submitted 2022-04-11; First posted 2022-06-15 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteer
MeSH Terms: interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capivasertib (Experimental): film-coated tablet, 200 mg
  Interventions: Drug: Capivasertib film-coated tablet, 200 mg
- [14C]AZD5363 (Capivasertib) (Experimental): Solution for Infusion 20 µg/mL (NMT 37.0 kBq/5 mL) and Oral Solution, 400 mg (NMT 4.8 MBq)
  Interventions: Drug: [14C]AZD5363 (Capivasertib)

INTERVENTIONS:
Drug: Capivasertib film-coated tablet, 200 mg — 400mg dose, oral, fasted
  Arms: Capivasertib
Drug: [14C]AZD5363 (Capivasertib) — Solution for Infusion 20 µg/mL (NMT 37.0 kBq/5 mL) - 100 µg; 5 mL, Intravenous
  Oral Solution, 400 mg (NMT 4.8 MBq) - 400mg; 100mL, oral, fasted
  Arms: [14C]AZD5363 (Capivasertib)

SUMMARY:
The Sponsor is developing the test medicine, Capivasertib, for the potential treatment of primary breast and prostate cancer. This two-part healthy volunteer study will try to identify the absolute bioavailability (amount of the test medicine that enters the blood stream), mass balance recovery (how much radioactivity can be recovered from the urine and faeces) and the rates and routes of elimination of the test medicine.

DETAILED DESCRIPTION:
The Sponsor is developing the test medicine, Capivasertib, for the potential treatment of primary breast and prostate cancer. Cancer is a condition where cells in a specific part of the body grow and reproduce uncontrollably, causing a growth called a tumour. The cancerous cells can invade and destroy surrounding healthy tissue, including organs. The four most common types of cancer within the UK are: breast, lung, prostate and bowel cancer. This two-part healthy volunteer study will try to identify the absolute bioavailability (amount of the test medicine that enters the blood stream), mass balance recovery (how much radioactivity can be recovered from the urine and faeces) and the rates and routes of elimination of the test medicine. Two out of three recipes of the test medicine are radiolabelled with carbon-14. 'Radiolabelled' means that the test medicine has a radioactive component (carbon-14) which helps us to track where the test medicine is in the body. This study will consist of two periods involving up to eight healthy male volunteers aged 30-65 and will take place at one non-NHS site. In Part 1, volunteers will receive a single dose of 2 non-radiolabelled oral tablets in the fasted state followed by an intravenous infusion (solution into the vein) of radiolabelled test medicine 1 hour 15 mins minutes later. Volunteers will be discharged from the clinical unit on Day 5. In Part 2, volunteers will receive a single oral dose of a radiolabelled oral solution in the fasted state. Volunteers will be discharged on Day 8, however may be required to remain at the clinical unit until Day 10 if the mass balance criteria have not been met by Day 8. Volunteers will receive a follow up phone call between Day 15 and Day 19. Volunteer's blood, urine and faeces will be taken throughout the study for analysis of the test medicine, radiation and for safety. Volunteers are expected to be involved in this study for approximately 9 weeks from screening to the follow-up call.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Must be willing and able to communicate and participate in the whole study.
* Healthy males aged 30 to 65 years inclusive at the time of signing informed consent.
* Must be vasectomised (at least 6 months prior to screening) and must agree to adhere to the contraception requirements of the study.
* Have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive as measured at screening.
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)
* Provision of signed, written and dated informed consent for optional genetic research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History of any clinically significant disease or disorder (e.g. cardiovascular, pulmonary, GI (including but not limited to refractory nausea and vomiting, malabsorption syndrome, chronic GI diseases, previous cholecystectomy, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib), liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment, skin abnormalities and glucose metabolism abnormalities) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the ADME of drugs.
* History of latent or chronic infections (e.g. tuberculosis, recurrent sinusitis, genital herpes, urinary tract infections) or at risk of infection (surgery, trauma or significant infection within previous 90 days, history of skin abscesses within previous 90 days).
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to capivasertib. Hay fever is allowed unless it is active
* Any known or suspected hypersensitivity or contraindication to the components of the study drug, capivasertib, judged to be clinically relevant by the investigator.
* History of severe COVID-19 (e.g. hospitalisation, extracorporeal membrane oxygenation, mechanically ventilated) in the last 6 months.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Any clinically significant abnormal findings in vital signs, at screening or pre-dose, as judged by the investigator.
* QTcF >450 msec or QT >500 msec or other clinically significant ECG abnormality, as judged by the investigator, at screening or pre-dose, or a history of additional risk factors for Torsades de Points (e.g. heart failure, hypokalaemia, family history of long QT syndrome), which in the opinion of the Investigator may put the volunteer at risk.
* Evidence of current SARS-CoV-2 infection within 2 weeks of first IMP administration.
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator
* Total bilirubin (TBL) ≥1.5×the ULN or ≥3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia)
* Clinically significant abnormal fasting blood glucose or triglycerides at screening.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), and human immunodeficiency virus (HIV) 1 and 2 antibody.
* Evidence of renal impairment at screening, as indicated by an estimated CLcr of <70 mL/min using the Cockcroft-Gault equation.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer. Note: subjects consented and screened, but not randomised in this study or a previous Phase I study, are not excluded.
* Subjects who report to have previously received capivasertib.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
* Subjects who have been administered IMP in an ADME study in the last 12 months.
* Plasma donation within 1 month of screening or any donation or loss (e.g. due to trauma or surgery) of >500 mL blood within the previous 3 months or 1350 mL of blood in 12 months prior to current study.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than 4 g of paracetamol/acetaminophen per day), herbal remedies, vitamins, and minerals during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life. COVID-19 vaccines are accepted concomitant medications. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no pharmacodynamic (PD) activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardise the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study
* Use of drugs which are strong inhibitors or inducers of CYP3A4 or drugs that are sensitive to inhibition of CYP3A4 within 2 weeks prior to the first administration of IMP
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks or 5 half-lives, whichever is longer, prior to the first administration of IMP.
* Known or suspected history of alcohol or drug abuse in the past 2 years or excessive intake of alcohol (>21 units per week [1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type]) or as judged by the investigator.
* A confirmed positive alcohol breath test at screening or admission.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 6 months prior to screening.
* A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
* Confirmed positive screen for drugs of abuse at screening or admission to the clinical unit.
* Excessive intake of caffeine-containing drinks or food (e.g. coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g. >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the clinical unit.
* Subjects with pregnant or lactating partners.
* Planned in-patient surgery, dental procedure or hospitalisation during the study.
* Involvement of any AstraZeneca AB, Quotient or study site employee or their close relatives.
* Subjects who are regularly exposed to the risk of COVID-19 infection as per of their daily life (e.g. health care professionals working in COVID-19 wards or at emergency departments).
* Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e. during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who cannot communicate reliably with the investigator.
* Vulnerable subjects, e.g. kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Failure to satisfy the investigator of fitness to participate for any other reason.

In addition, the following is considered a criterion for the exclusion from the optional genetic component of the study:

- Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) | Plasma sample collection from pre-dose to 72 hours post dose
  Absolute bioavailability (F) of oral capivasertib compared to [14C]-capivasertib (part 1)
tmax | Plasma sample collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (part 1)
Cmax | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (part 1)
AUC0-t | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (Part 1)
AUC0-inf | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (Part 1)
t1/2 | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (Part 1)
λz | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (Part 1)
CL/F | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (Part 1)
Vz/F | Plasma samples collection from pre-dose to 72 hours post dose
  PK of capivasertib and [14C]AZD5363 (capivasertib) in plasma (Part 1)
tmax | Plasma sample collection from pre-dose to 168 hours post dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
Cmax | Plasma sample collection from pre-dose to 168 hours post dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
AUC0-t | Plasma sample collection from pre-dose to 168 hours post dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
AUC0-inf | Plasma sample collection from pre-dose until 168 hours post-dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
t1/2 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
λz | Plasma sample collection from pre-dose until 168 hours post-dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
CL/F | Plasma sample collection from pre-dose until 168 hours post-dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
Vz/F | Plasma sample collection from pre-dose until 168 hours post-dose
  PK (plasma) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
CLR | Plasma sample collection from pre-dose to 72 hours post dose and urine samples collected from pre-dose until 168 hours post-dose
  PK (plasma and urine) and total radioactivity (whole blood and plasma) of capivasertib (Part 2)
CumAe | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of [14C]AZD5365 (capivasertib) from urine and faecal samples (Part 2)
Cum%Ae | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of [14C]AZD5365 (capivasertib) from urine and faecal samples (Part 2)
Ae | Urine and faecal sample collection from pre-dose until 168 hours post-dose
  Mass balance recovery of [14C]AZD5365 (capivasertib) from urine and faecal samples (Part 2)
%Ae | Urine and faecal sample collection from pre-dose until 168 hours post-dose
  Mass balance recovery of [14C]AZD5365 (capivasertib) from urine and faecal samples (Part 2)
Blood:plasma concentration ratios | Whole blood samples collected up to 24 hours post dose. Plasma sample collection from pre-dose until 72 hours post-dose
  Blood:plasma concentration ratios of total radioactivity (Part 2)

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events | Through study duration, an average of 9 weeks.
  To provide additional safety and tolerability information for capivasertib by assessing the incidence of AEs (Part 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom